CLINICAL TRIAL: NCT05437445
Title: Utilizing Augmented Artificial Intelligence for Aminoacidopathies: Experience of Collaborative Laboratory Integrated Reporting From Pakistan
Brief Title: Utilizing Augmented Artificial Intelligence for Aminoacidopathies
Status: Completed | Type: Observational
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Zaib Un Nisa Khan, PRINCIPAL INVESTIGATOR, Aga Khan University Hospital, Pakistan
Other Study IDs: ERC # 2019-1709-4536
Record Dates: First submitted 2022-06-25; First posted 2022-06-29 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Inborn Errors of Metabolism
Keywords: Clinical Laboratory Integrated Reports (CLIR); Inherited metabolic disorders (IMDs)
MeSH Terms: conditions — Metabolism, Inborn Errors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases Data: subjects having abnormal plasma amino acid profiles with either one or more amino acid concentrations beyond (high or low) the locally defined age-specific reference ranges
  Interventions: Diagnostic Test: Plasma amino acid assay

INTERVENTIONS:
Diagnostic Test: Plasma amino acid assay — Plasma amino acid analysis was performed on all the blood samples received in biogenetics lab at Aga khan university, Karachi during one year period.

SUMMARY:
The objective of the study was to interpret metabolic profiles of plasma amino acid (PAA) and compare reference intervals (RI) of PAA data from Pakistan with data from other countries using Clinical Laboratory Integrated Reports (CLIR). One-year data (reference and cases data) of twenty-two PAA, analyzed by ion exchange high performance chromatography at Biochemical Genetics Laboratory (BGL) of Aga Khan University Pakistan, was compiled in a comma-separated values (.csv) file and uploaded on CLIR Software using AAQP (Amino Acid in Plasma) application for statistical analysis. Among total of 2081 PAA profiles, 92% (n=1913) were completely normal with all PAA values falling within the age-specific reference range. A concordance of 98.8% was noted between the reporting done by the BGL at AKU and then after applying CLIR tools.

ELIGIBILITY:
Inclusion Criteria:

All plasma samples during 1 year received at Biogenetic Lab

Exclusion Criteria:

Subjects with age greater than 16 years

Ages: 1 Year to 16 Years | Sex: All
Age Groups: Child
Study Population: Data of all those who had Plasma amino acid analyzed at the Biogenetic laboratory of Aga Khan University, symptomatic as well as asymptomatic children with suspicion of Inherited Metabolic Disorders (IMDs), from August 2019-August 2020 were included. Plasma amino acids analysis was performed using cation-exchange high-performance liquid chromatography (HPLC) on Biochrom 30+ model using lithium column diameter 4.6 mm and detected at 440/570 nm.
Sampling Method: Non-Probability Sample
Enrollment: 2081 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
postanalytical interpretation of concentration of plasma leucin, isoleucine and valine in nmol/L using Clinical Laboratory Integrated Reports (CLIR) | 1 year
  Clinical Laboratory Integrated Reports (CLIR, formerly Region 4 Stork) is a post-analytical software that compares the amino acid results against a large database of reference ranges, disease-specific cutoffs, and ratios of diagnostic markers. Among 168 subjects having abnormal PAA profiles in our lab, 10.1% were correctly classified as MSUD and 100% concordance with CLIR reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Dr lena Jafri, Principal Investigator — Aga khan hospital karachi, Pakistan
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No